CLINICAL TRIAL: NCT00670020
Title: Supplemental Perioperative Oxygen to Reduce the Incidence of Post-Cesarean Endometritis and Wound Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Carolyn Gardella, MD, MPH, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18821
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Wound Infection or Endometritis Post Cesarean Section
Keywords: Women undergoing Cesarean section after the onset of labor
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): supplemental perioperative oxygen
  Interventions: Procedure: supplemental perioperative oxygen
- 2 (No Intervention): Normal

INTERVENTIONS:
Procedure: supplemental perioperative oxygen — increased perioperative oxygen verses non-interventional oxygen
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether supplemental perioperative oxygen significantly decreases the incidence of post-Cesarean endometritis and wound infection among women who undergo Cesarean section after the onset of labor.

DETAILED DESCRIPTION:
Women undergoing cesarean section after rupture of membranes or onset of labor are randomized in a one to one ratio to either normal or supplemental perioperative oxygen during cesarean section and for two hours afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent a clinically indicated cesarean delivery after the onset of labor or rupture of membranes

Exclusion Criteria:

* Cesarean delivery prior to the onset of labor or rupture of membranes
* emergent cesarean delivery
* general endotracheal anesthesia
* clinical chorioamnionitis
* HIV infection
* less than 16 years of age

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2001-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
surgical site infection | within two weeks of cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Gardella, MD, MPH, Principal Investigator — University of Washington Dept of Ob/Gyn